CLINICAL TRIAL: NCT03905213
Title: Impact of the Use of Three Dressings in the Prevention of Surgical Wound Infection in Patients Undergoing Mayor Cardiac Surgery: a Clinical Prospective and Randomized Study
Brief Title: Prevention of Surgical Wound Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Jesus Perez (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Maria Jesus Perez, Principal Investigator, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MICRO.HGUGM.2018-008
Record Dates: First submitted 2019-03-20; First posted 2019-04-05 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-03

CONDITIONS: Cardiac Surgery

STUDY DESIGN:
Intervention Model Description: randomized in three groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional gauze (Active Comparator): Device is a conventional gauze and the change will be to the day 2 and 4 of surgery
  Interventions: Device: dressing MEPORE
- polyurethane dressing (Experimental): Device is a polyurethane dressing and the change will be to the day 7 of surgery
  Interventions: Device: dressing MEPILEX
- vacuum therapy dressing (Experimental): Device is a vacuum therapy dressing and the change will be to the day 7 of surgery
  Interventions: Device: dressing PICCO

INTERVENTIONS:
Device: dressing MEPORE — assignation to three different authorised and on label dressing: conventional dressing (MEPORE)
  Arms: conventional gauze
Device: dressing MEPILEX — assignation to three different authorised and on label dressing: absorbent(MEPILEX)
  Arms: polyurethane dressing
Device: dressing PICCO — assignation to three different authorised and on label dressing:vacuum Therapy dressing(PICCO)
  Arms: vacuum therapy dressing

SUMMARY:
To compare cost effectiveness of a polyurethane dressing or a vacuum therapy dressing versus the conventional gauze in the prevention of superficial wound infection y major cardiac surgery

DETAILED DESCRIPTION:
It is a clinical prospective and randomized study. patientes will be randomized to three groups on the day of surgery: conventional gauze, polyurethane or vacuum therapy dressing. Clinical al microbiological data will be monitorized to evaluate the infection rate of surgical wound , mediastinitis, days of hospital stay and consumption of antimicrobials.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled to cardiac surgery.
* signed informed consent form

Exclusion Criteria:

* hypersensibility to dressings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-08-28 (Estimated); Study Completion 2021-08-28 (Estimated)

PRIMARY OUTCOMES:
prevention of surgical wound infection | surgery date up to 6 months
  surgical wound infection measured as number of patients suffering surgical wound infection during the study period

SECONDARY OUTCOMES:
hospital stay | from hospitalization until an average of 1 year
  days at hospital
antimicrobial consumption | from surgery date until an average of 1 year
  defined dose of antimicrobial agents during hospital stay
dressing consumption cost | from surgery date until an average of 8 weeks
  number of dressing and its cost

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus Perez Granda, PhD, Principal Investigator — Gregorio Marañón Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perez-Granda MJ, Cuerpo G, Barrio JM, Valerio M, Munoz P, Pinto AG, Valencia DE, Vicario FS, Bouza E; Cardiovascular Infection Study Group. A prospective randomized study that compares three different dressings for the prevention of surgical site infections following major heart surgery. Sci Rep. 2025 Jun 6;15(1):19960. doi: 10.1038/s41598-025-02533-7. PMID 40481025